CLINICAL TRIAL: NCT03684330
Title: Efficacy of Vitamin D Supplementation Added to WBV Chronic Protocol in Inflammatory Markers, Peripheral and Respiratory Strength and Body Composition in Old Patients With COPD
Brief Title: Vitamin D Supplementation and WBV in Inflammatory Markers, Strength and Body Composition in Old Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maíra F Pessoa (Other)
Responsible Party: Sponsor-Investigator, Maíra F Pessoa, Clinical Professor, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: croninflam
Record Dates: First submitted 2018-09-22; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: COPD; Aging
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplementation (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D; Other: whole body vibration (WBV)
- Vitamin D placebo (Placebo Comparator)
  Interventions: Other: whole body vibration (WBV)

INTERVENTIONS:
Dietary Supplement: Vitamin D — a dose once a week
  Arms: Vitamin D supplementation
Other: whole body vibration (WBV) — 03 months of WBV training three times per week

SUMMARY:
Verify the influence off vitamin D supplementation and a whole body vibration (WBV) protocol during 03 months in older patients chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* Older patients with COPD
* Both genders
* Sedentary according to International Physical Activity Questionnaire (IPAQ) short form
* BMI in between 22.9 and 28 kg/m2.
* Older patients with COPD should have a clinical-functional diagnosis of the disease according to GOLD (GOLD, 2018), have been ex-smokers and have not used corticosteroids or have used this drug in a stable way for at least one year (without dosage or medication modifications).
* Older volunteers should be self-referenced healthy or, if they had systemic arterial hypertension or diabetes mellitus, these comorbidities should be controlled by diet or regular medication use.

Exclusion Criteria:

* Older patients with COPD who had episodes of exacerbation in the last three months, those with pulmonary rehabilitation programs in the last year, those who used home oxygen therapy, and patients with COPD associated comorbidities were excluded.
* Volunteers of both groups who were taking vitamin D were excluded, as well as the current smokers, although occasional, volunteers with a history of labyrinthitis or thromboembolism, who had undergone surgical procedures of any size in the last year, such as plaques, pins or cardiac pacemakers, those with unconsolidated fractures that used medications that affected bone metabolism or lean mass, or those who had difficulties adapting to the assessment or the training protocol.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
serum inflammatory marker Interleukine-6 (IL-6) | before and immediately up to 12 weeks in WBV training.
  changes in total serum values of interleukine 6
serum inflammatory marker Interleukine-8 (IL-8) | before and immediately up to 12 weeks in WBV training.
  changes in total serum values of interleukine 8
serum inflammatory marker TNF-alpha ( and BDNF) | before and immediately up to 12 weeks in WBV training.
  changes in total serum values of tumoral necrose factor alpha
serum inflammatory marker and brain derived neurotrophic factor (BDNF) | before and immediately up to 12 weeks in WBV training.
  changes in total serum values of brain derived neurotrophic factor

SECONDARY OUTCOMES:
Peripheral strength | before and immediately up to 12 weeks in WBV training.
  Changes in Peripheral muscle strength assessed by the hand dynamometer (device that assess strength) in values obtained from the mean of 03 maneuvers of isokinetic contraction, in centimeters of water
Body composition | before and immediately up to 12 weeks in WBV training.
  Changes in electrical bioimpedance assessing lean mass in segmental areas and trunk
Respiratory strength | before and immediately up to 12 weeks in WBV training.
  Changes in respiratory strength obtained from a manovacuometer, collecting the major value of 03 maneuvers of the maximal inspiration (vacuometer) to the maximal expiration pressures (manometer), with values obtained in centimeters of water

CONTACTS AND LOCATIONS:
Locations (1):
- UFPE, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided